CLINICAL TRIAL: NCT07126717
Title: Confirmatory Study on the Acute Effects of Zynamite® S on Cognitive Function and Mood in University Students: a Randomized, Double-blind, Placebo-controlled Crossover Study
Brief Title: Acute Effects of Zynamite® S in Cognitive Function and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nektium Pharma SL (Industry)
Collaborators: University of Atlántico Medio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYNS_HCT_2025.01
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Performance; Mood
Keywords: Zynamite® S; Mango Leaf Extract; Cognitive Performance; Mood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Capsule containing food-grade maltodextrin
  Interventions: Dietary Supplement: Placebo
- Zynamite® S 100mg (Experimental): Capsule containing 100 mg of soluble mango leaf extract (Zynamite® S) standardized to 60% of mangiferin
  Interventions: Dietary Supplement: Zynamite® S

INTERVENTIONS:
Dietary Supplement: Placebo — Food-grade maltodextrin
  Arms: Placebo
Dietary Supplement: Zynamite® S — Water-soluble mango leaf extract standardized to 60% of mangiferin
  Arms: Zynamite® S 100mg

SUMMARY:
The present study sought to confirm the cognitive and mood benefits of a standardized soluble mango leaf extract, named as Zynamite® S. A placebo or a single dose of the botanical extract (100 mg) was administered and its acute effects on mental function and mood were evaluated before product intake, at 30 min, 3 h, and 5 h post-ingestion.

DETAILED DESCRIPTION:
The present study is a double-blind, randomized, placebo-controlled crossover clinical trial that aimed to evaluate the effects of a standardized soluble mango leaf extract (Zynamite® S) on cognitive performance and mood. The study included 88 healthy university students aged 18-25 years. Participants received a single 100 mg dose of Zynamite® S or a placebo. Cognitive performance was evaluated by using the Trail Making Test (TMT) to assess executive functions, the Digit Symbol Substitution Test (DSST) for processing speed, and the Stroop Color and Word Test and the Stroop Interference Test to evaluate selective attention and cognitive flexibility. Additionally, mood was assessed using the Spanish short version of the Profile of Mood States (POMS). All the assessments were conducted before product intake, at 30 min, 3 h, and 5 h post-ingestion.

ELIGIBILITY:
Inclusion Criteria:

* Being registered as an undergraduate or postgraduate university student
* Being between 18 and 25 years old
* Being healthy and free of any relevant medical condition or illness

Exclusion Criteria:

* Suffering from chronic diseases such as asthma, type 1 diabetes, thyroid diseases (such as hypothyroidism or hyperthyroidism), autoimmune disorders (such as Crohn's disease), and psychiatric conditions such as anxiety disorders, major depression, eating disorders (anorexia, bulimia), attention deficit hyperactivity disorder (ADHD), among others
* Being pregnant or lactating
* Having any known intolerance, hypersensitivity, or allergies to any of the ingredients of the investigational products
* Having intestinal malabsorption problems, as well as learning difficulties, dyslexia, eye problems, or color blindness
* Intaking of psychoactive substances or medications that could influence the study results, such as consuming >500 mg of caffeine per day (>6 cups of 150 ml filtered coffee) and/or alcohol
* Having comprehension or communication difficulties that prevent full understanding of the informed consent or effective participation in the study, such as autism spectrum disorders, aphasia, or intellectual disability

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Changes in Trail Making Test (TMT) Score | At baseline (30 minutes before supplement intake), at 30 minutes, 3 hours, and 5 hours after supplement intake.
  Changes in the Trail Making Test (TMT) score will be used to evaluate executive functions between placeobo and Zynamite® S groups.
  This test is divided into two parts wtih 25 items each: Part A (TMT-A), which evaluates psychomotor attention and speed and involves connecting consecutively numbered circles, and Part B (TMT-B), which requires connecting alternating circles of letters and numbers and is used to measure executive function. A longer time taken to complete the test is interpreted as poorer performance.
Changes in Digit symbol substitution test (DSST) Score | At baseline (30 minutes before supplement intake), at 30 minutes, 3 hours, and 5 hours after supplement intake.
  Changes in the Digit symbol substitution test (DSST) will be employed to compare performance on processing speed, attention, and working memory between placebo and Zynamite® S groups.
  DSST is a paper-and-pencil cognitive test presented on a single sheet of paper, requiring the subject to match symbols with numbers according to a key located at the top of the page. The subject copies the symbol into spaces beneath a row of numbers. The score is based on the number of correct symbols the participant manages to substitute within 90 s.
Changes in Stroop Color and Word & Stroop Interference Score | At baseline (30 minutes before supplement intake), at 30 minutes, 3 hours, and 5 hours after supplement intake.
  Changes in the Stroop Color and Word Test and Stroop Interefernce Test will be used to assess cognitive functions, such as selective attention and cognitive flexibility between placebo and Zynamite® S groups.
  The Stroop Color and Word Test consists on three 45-second tasks. First, the participants read color words printed in black ink (the 'P' score). Next, they name the ink color of "XXXX" symbols (the 'C' score). In the final interference stage, the participant must state the ink color of a word that is printed in a conflicting color, such as the word "BLUE" printed in red ink (the 'PC' score). These three scores are then used to calculate a final T score of interference, where a higher score indicates better performance and attention control.

SECONDARY OUTCOMES:
Changes in Profile of Mood States (POMS) Score | At baseline (30 minutes before supplement intake), at 30 minutes, 3 hours, and 5 hours after supplement intake.
  Changes on the Profile of Mood States (POMS) score will be used to evaluate mood and well-being between placebo and Zynamite® S groups.
  Participants will complete the Spanish short version of the POMS 65-item questionnaire, which includes a total of 6 subscales: tension (score range 0 to 36), depression (score range 0 to 60), anger (score range 0 to 48), fatigue (score range 0 to 28), vigor (score range 0 to 32), and confusion (score range 0 to 28), as well as a total mood disturbance score (score range -32 to 200). The total mood disturbance score is calculated by summing the five negative subscale scores (tension, depression, anger, fatigue, and confusion) and subtracting the vigor score. Higher scores for the total mood disturbance indicate a greater degree of mood disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Atlántico Medio, Tafira Baja, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellote-Caballero Y, Beltran-Arranz A, Aibar-Almazan A, Carcelen-Fraile MDC, Rivas-Campo Y, Lopez-Rios L, Vega-Morales T, Gonzalez-Martin AM. Acute Supplementation of Soluble Mango Leaf Extract (Zynamite(R) S) Improves Mental Performance and Mood: A Randomized, Double-Blind, Placebo-Controlled Crossover Study. Pharmaceuticals (Basel). 2025 Apr 14;18(4):571. doi: 10.3390/ph18040571. PMID 40284006
- [Background] Fuentes-Rios D, Sanchez-Rodriguez A, Lopez-Rios L, Garcia-Gonzalez E, Martinez-Canton M, Galvan-Alvarez V, Gallego-Selles A, Martin-Rincon M, Calbet JAL, Vega-Morales T. Human Pharmacokinetic Profiling and Comparative Analysis of Mangiferin and Its Monosodium Derivative from Mangifera indica Extracts Using UHPLC-MS/MS with 1H NMR and MALDI-TOF Confirmation. Molecules. 2025 Jan 21;30(3):461. doi: 10.3390/molecules30030461. PMID 39942566
- [Background] Sharif S, Guirguis A, Fergus S, Schifano F. The Use and Impact of Cognitive Enhancers among University Students: A Systematic Review. Brain Sci. 2021 Mar 10;11(3):355. doi: 10.3390/brainsci11030355. PMID 33802176
- [Background] Malik M, Tlustos P. Nootropics as Cognitive Enhancers: Types, Dosage and Side Effects of Smart Drugs. Nutrients. 2022 Aug 17;14(16):3367. doi: 10.3390/nu14163367. PMID 36014874
- [Background] Jangra A, Lukhi MM, Sulakhiya K, Baruah CC, Lahkar M. Protective effect of mangiferin against lipopolysaccharide-induced depressive and anxiety-like behaviour in mice. Eur J Pharmacol. 2014 Oct 5;740:337-45. doi: 10.1016/j.ejphar.2014.07.031. Epub 2014 Jul 23. PMID 25064341
- [Background] Cao C, Su M, Zhou F. Mangiferin inhibits hippocampal NLRP3 inflammasome and exerts antidepressant effects in a chronic mild stress mice model. Behav Pharmacol. 2017 Aug;28(5):356-364. doi: 10.1097/FBP.0000000000000305. PMID 28410265
- [Background] Lum PT, Sekar M, Gan SH, Pandy V, Bonam SR. Protective effect of mangiferin on memory impairment: A systematic review. Saudi J Biol Sci. 2021 Jan;28(1):917-927. doi: 10.1016/j.sjbs.2020.11.037. Epub 2020 Nov 13. PMID 33424383
- [Background] Lei LY, Wang RC, Pan YL, Yue ZG, Zhou R, Xie P, Tang ZS. Mangiferin inhibited neuroinflammation through regulating microglial polarization and suppressing NF-kappaB, NLRP3 pathway. Chin J Nat Med. 2021 Feb;19(2):112-119. doi: 10.1016/S1875-5364(21)60012-2. PMID 33641782
- [Background] Li HW, Lan TJ, Yun CX, Yang KD, Du ZC, Luo XF, Hao EW, Deng JG. Mangiferin exerts neuroprotective activity against lead-induced toxicity and oxidative stress via Nrf2 pathway. Chin Herb Med. 2019 Dec 14;12(1):36-46. doi: 10.1016/j.chmed.2019.12.002. eCollection 2020 Jan. PMID 36117559
- [Background] Alberdi E, Sanchez-Gomez MV, Ruiz A, Cavaliere F, Ortiz-Sanz C, Quintela-Lopez T, Capetillo-Zarate E, Sole-Domenech S, Matute C. Mangiferin and Morin Attenuate Oxidative Stress, Mitochondrial Dysfunction, and Neurocytotoxicity, Induced by Amyloid Beta Oligomers. Oxid Med Cell Longev. 2018 Jun 14;2018:2856063. doi: 10.1155/2018/2856063. eCollection 2018. PMID 30013719
- [Background] Lopez-Rios L, Wiebe JC, Vega-Morales T, Gericke N. Central nervous system activities of extract Mangifera indica L. J Ethnopharmacol. 2020 Oct 5;260:112996. doi: 10.1016/j.jep.2020.112996. Epub 2020 May 27. PMID 32473365
- [Background] Wightman EL, Jackson PA, Forster J, Khan J, Wiebe JC, Gericke N, Kennedy DO. Acute Effects of a Polyphenol-Rich Leaf Extract of Mangifera indica L. (Zynamite) on Cognitive Function in Healthy Adults: A Double-Blind, Placebo-Controlled Crossover Study. Nutrients. 2020 Jul 23;12(8):2194. doi: 10.3390/nu12082194. PMID 32717999